CLINICAL TRIAL: NCT06821191
Title: Comparison of Dual Antiplatelet Therapy De-escalation by Dose Reduction Versus Switching in Patients Undergoing PCI: A Prospective, Randomized Pharmacodynamic Study - The Switching Antiplatelet-8 (SWAP-8) Study
Brief Title: Comparison of Dual Antiplatelet Therapy De-escalation by Dose Reduction Versus Switching in Patients Undergoing PCI: The Switching Antiplatelet-8 (SWAP-8) Study
Acronym: SWAP-8
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202401735
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; DAPT de-escalation; DAPT; dose-reduction; switch; clopidogrel; prasugrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Intervention Model Description: The proposed investigation will be a prospective, randomized, parallel-design, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DAPT de-escalation by switch (Active Comparator)
  Interventions: Drug: clopidogrel 75 mg
- DAPT de-escalation by dose-reduction (Experimental)
  Interventions: Drug: Prasugrel 5 mg

INTERVENTIONS:
Drug: clopidogrel 75 mg — Clopidogrel 75 mg od for 30 ± 5 days
  Arms: DAPT de-escalation by switch
Drug: Prasugrel 5 mg — Prasugrel 5 mg od for 30 ± 5 days
  Arms: DAPT de-escalation by dose-reduction

SUMMARY:
Dual antiplatelet therapy (DAPT) with low-dose aspirin and a P2Y12 inhibitor is the current standard of care in patients with coronary artery disease experiencing an acute event or undergoing percutaneous coronary intervention. However, the ischemic benefits are counterbalanced by a significant increase in bleeding events. Over time, different DAPT de-escalation strategies have been developed to reduce the bleeding risk while maintaining the ischemic protection, but there is currently no head-to-head comparison between them. The purpose of this clinical trial is to conduct a head-to-head comparison on the pharmacodynamic efficacy of DAPT de-escalation by dose reduction to low-dose prasugrel (5 mg od) and DAPT de-escation by switching from standard-dose more potent P2Y12 receptor inhibitor to standard-dose clopidogrel (75 mg). To determine if the PD profiles of these two strategies are comparable, we aim to conduct a non-inferiority study.

DETAILED DESCRIPTION:
The combination of low-dose aspirin and a P2Y12 receptor inhibitor, commonly referred as dual antiplatelet therapy (DAPT), is guideline-recommended for preventing atherothrombotic events in patients experiencing an acute coronary syndrome (ACS) or undergoing percutaneous coronary intervention (PCI). In ACS patients undergoing PCI, DAPT is initiated at the time of the event and maintained for up to one year to mitigate the risks of stent-related complications and ischemic recurrences.4 There are 3 currently available oral P2Y12 inhibitors: clopidogrel, prasugrel, and ticagrelor. Among ACS patients undergoing PCI, prasugrel and ticagrelor are recommended over clopidogrel because of their enhanced efficacy in reducing ischemic events, including stent thrombosis. However, the increased antiplatelet potency of prasugrel and ticagrelor enhances the risk of bleeding, which has detrimental effects on the overall patient prognosis. The increased risk of mortality in patients experiencing bleeding events underscores the need for antiplatelet strategies that reduce bleeding risk while maintaining significant ischemic protection.

The majority of recurrent ischemic events, including stent thrombosis, tend to occur within the first 1 to 3 months after the index PCI procedure. As a result, in clinical practice it is common to use more potent antiplatelet therapies during the early (i.e., 1-3) months post-PCI, when platelet reactivity is heightened, and transition to therapies with lower platelet inhibition thereafter. This strategy, aimed at reducing bleeding risks while providing ischemic protections, is referred to as de-escalation and its implementation is supported by practice guidelines. In line with Academic Research Consortium (ARC) definitions, de-escalation can be implemented in 3 ways: a) by switching from a more potent to a less potent P2Y12 inhibitor; b) by dose reduction (e.g., lowering prasugrel or ticagrelor doses as an alternative to the initial regimen) or c) by stopping one antiplatelet drug (e.g., either the P2Y12 inhibitor or aspirin). Of the available de-escalation strategies, two of these allow patients to remain on a DAPT regimen maintaining the synergistic effect of targeting two different platelet activation pathways: de-escalation by switch and de-escalation by dose reduction. Notably, pharmacodynamic (PD) response to clopidogrel is characterized by a significant interindividual variability, which is partially mediated by specific alleles encoding the cytochrome P450 2C19. Thus, carriers of these alleles may be at increased risk of thrombotic events if a DAPT de-escalation by switch to clopdogrel is pursued.

In contrast, de-escalation by dose reduction has limited supporting evidence and low adoption in clinical practice. With a de-escalation by dose reduction strategy, patients remain on a potent P2Y12 inhibitor (i.e., prasugrel or ticagrelor) but at lower doses, which can reduce side effects, such as bleeding, without compromising efficacy, as these drugs have a more predictable PD response compared to clopidogrel. To date, clinical trial data on dose reduction after the early acute phase (i.e., 1-3 months) in patients with ACS undergoing PCI is limited and shown only with prasugrel. Notably, a recent head-to-head randomized controlled trial favoring prasugrel over ticagrelor, along with the availability of generic formulations of prasugrel, has led to a shift in antiplatelet prescriptions toward prasugrel. However, although there is extensive evidence comparing various de-escalation strategies with standard-of-care DAPT regimens, there are very few studies directly comparing de-escalation strategies with each other, setting the rationale for this investigation. To determine if the pharmcodynamic profiles of DAPT de-escalation by dose-reduction and by switching to clopidogrel are comparable, we aim to conduct a non-inferiority study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone PCI and are on maintenance treatment with DAPT, consisting of low-dose aspirin with either prasugrel (10 mg qd) or ticagrelor (90 mg bid) as part of standard of care. In particular, patients who underwent PCI in the setting of an acute coronary syndrome will be eligible for randomization after ≥90 days post-PCI, while patients who underwent PCI in the setting of a chronic coronary syndrome ≥30 days post-PCI.
2. Age ≥18 years.
3. Provide written informed consent.

Exclusion Criteria:

1. Prior history of stent thrombosis
2. Prior cerebrovascular event
3. PCI within 30 days
4. Predicted poor metabolizer of clopidogrel based on CYP2C19 genotyping (e.g., *2/*2 or *3/*3),
5. On treatment with any oral anticoagulant (vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxaban) or chronic low-molecular-weight heparin (at venous thrombosis treatment, not for prophylaxis)
6. Hemodynamic instability
7. Hypersensitivity to Aspirin, Clopidogrel, or Prasugrel
8. Known hematologic malignancies or thrombocytopenia (platelet count <80x106/mL)
9. Known hemoglobinopathies or anemia (hemoglobin <9 g/dL)
10. Pregnant and breastfeeding women [women of childbearing age must use reliable birth control (i.e., oral contraceptives) while participating in the study].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Platelet reactivity measured by VerifyNow | 30±5 days
  The primary endpoint of the study will be to establish non-inferiority by comparing PRU levels, determined using the VerifyNow system, between de-escalation through dose reduction to low-dose prasugrel (5 mg qd) and de-escalation through switching to standard-dose clopidogrel (75 mg qd) at trough levels.

SECONDARY OUTCOMES:
Platelet reactivity measured by VerifyNow | 30±5 days
  If non-inferiority is established, a superiority analysis will be conducted by comparing PRU levels, determined using the VerifyNow system, between de-escalation through dose reduction to low-dose prasugrel (5 mg qd) and de-escalation through switching to standard-dose clopidogrel (75 mg qd) at trough levels.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erlinge D, Ten Berg J, Foley D, Angiolillo DJ, Wagner H, Brown PB, Zhou C, Luo J, Jakubowski JA, Moser B, Small DS, Bergmeijer T, James S, Winters KJ. Reduction in platelet reactivity with prasugrel 5 mg in low-body-weight patients is noninferior to prasugrel 10 mg in higher-body-weight patients: results from the FEATHER trial. J Am Coll Cardiol. 2012 Nov 13;60(20):2032-40. doi: 10.1016/j.jacc.2012.08.964. Epub 2012 Oct 17. PMID 23083774
- [Background] Erlinge D, Gurbel PA, James S, Lindahl TL, Svensson P, Ten Berg JM, Foley DP, Wagner H, Brown PB, Luo J, Zhou C, Moser BA, Jakubowski JA, Small DS, Winters KJ, Angiolillo DJ. Prasugrel 5 mg in the very elderly attenuates platelet inhibition but maintains noninferiority to prasugrel 10 mg in nonelderly patients: the GENERATIONS trial, a pharmacodynamic and pharmacokinetic study in stable coronary artery disease patients. J Am Coll Cardiol. 2013 Aug 13;62(7):577-83. doi: 10.1016/j.jacc.2013.05.023. Epub 2013 Jun 7. PMID 23747759
- [Background] Capodanno D, Mehran R, Krucoff MW, Baber U, Bhatt DL, Capranzano P, Collet JP, Cuisset T, De Luca G, De Luca L, Farb A, Franchi F, Gibson CM, Hahn JY, Hong MK, James S, Kastrati A, Kimura T, Lemos PA, Lopes RD, Magee A, Matsumura R, Mochizuki S, O'Donoghue ML, Pereira NL, Rao SV, Rollini F, Shirai Y, Sibbing D, Smits PC, Steg PG, Storey RF, Ten Berg J, Valgimigli M, Vranckx P, Watanabe H, Windecker S, Serruys PW, Yeh RW, Morice MC, Angiolillo DJ. Defining Strategies of Modulation of Antiplatelet Therapy in Patients With Coronary Artery Disease: A Consensus Document from the Academic Research Consortium. Circulation. 2023 Jun 20;147(25):1933-1944. doi: 10.1161/CIRCULATIONAHA.123.064473. Epub 2023 Jun 19. PMID 37335828